CLINICAL TRIAL: NCT05320211
Title: Three-dimensional Printed Orthoses for Improving Daily Functioning in Chronic Hand Conditions
Brief Title: Three-dimensional Printed Hand Orthoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Merel Brehm, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10310012110002
Record Dates: First submitted 2022-03-24; First posted 2022-04-11 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Hand Injuries and Disorders
Keywords: feasibility; hand; orthotic device; printing; three-dimensional; activities, daily living; satisfaction; production time; costs
MeSH Terms: conditions — Hand Injuries; Disease; Motor Activity; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: within-subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D-printed hand orthoses (Experimental)
  Interventions: Device: 3D-printed hand orthosis

INTERVENTIONS:
Device: 3D-printed hand orthosis — 3D-printed hand orthoses (intervention) will be compared with custom-fabricated conventional orthoses (control condition at baseline)

SUMMARY:
In persons with chronic hand conditions, orthoses are often prescribed to improve daily-life functioning. In most cases, orthoses are custom manufactured based on a plaster hand model, which is a time-consuming and labor-intensive process. It has been demonstrated that the production time to custom manufacture hand orthoses can be greatly reduced by using three-dimensional (3D) scanning and printing, offering a promising cost-effective alternative to conventional costum manufactured hand orthoses. However, before setting up a cost-effectiveness study in persons with chronic hand conditions, insight into the effectiveness of 3D-printed orthoses on performance of activities of daily living (ADL) is needed, as well as insight into potential cost reductions. To date, this information is largely unknown. The aims of this feasibility study are 1) to collect data on the preliminary effectiveness of 3D-printed orthoses on performance of ADL, satisfaction with the orthosis and quality of life compared to conventional orthoses in persons with chronic hand conditions, and 2) to compare the production time and costs of 3D-printed orthoses with conventional orthoses.

ELIGIBILITY:
Inclusion Criteria:

1. Having a chronic hand-wrist condition due to an injury, or a musculoskeletal disorder, neuromuscular disorder, or neurological disorder;
2. Minimum age of 18 years;
3. Currently wearing a conventional custom manufactured hand orthosis (including a wrist-orthosis, wrist/thumb orthosis or thumb orthosis) for permanent use;
4. Indicated for a new hand orthosis.

Exclusion Criteria:

1. Already wearing a 3D-printed orthosis
2. Wearing a silver wrist-orthosis, wrist/thumb orthosis or thumb orthosis
3. Wearing an orthosis prescribed for a dysfunctional hand;
4. Wearing a broken orthosis;
5. Wearing the orthosis only at night;
6. Worsening of disease;
7. Insufficient mastery of the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in performance of ADL on the custom short form of the Dutch-Flemish Patient-Reported Outcomes Measurement Information System - Upper extremity (DF-PROMIS-UE) at 4 months post-intervention. | 2 weeks pre-intervention; baseline; 1 month post-intervention; 4 months post-intervention
  The short form DF-PROMIS-UE contains 25 items from the DF-PROMIS-UE 46-item bank. Patients will rate how easily they can perform each activity on a 5-point scale, ranging from "without any difficulty" (score 4 or 5) to "unable to do" (score 1). For each activity, the question was added whether participants use their orthosis for that specific activity. The total score will be expressed as a T-score, which is a standardized score, with 50 representing the average score of the US general population and 10 being its standard deviation (SD). Note. For this study, the reliability of the DF-PROMIS-UE in persons with chronic hand conditions will be determined.

SECONDARY OUTCOMES:
Change from baseline in performance of ADL, overall hand function, pain, work, performance, aesthetics, and satisfaction on the Michigan Hand Questionnaire-Dutch Language version (MHQ-DLV) at 4 months post-intervention. | 2 weeks pre-intervention; baseline; 1 month post-intervention; 4 months post-intervention
  MHQ-DVL domain items are scored from 0 - 100, in which 100 is the best possible ability, while for pain a score of 0 indicates no pain. The total MHQ-DLV score is calculated as the mean of all 6 domains (after converting pain from a "best score of 0" scale to a "best score of 100" scale). Note. For this study, the reliability of the MHQ-DLV in persons with chronic hand conditions will be determined.
Change from baseline in satisfaction assessed with the Dutch version of the Client Satisfaction with Device (CSD) module of the Orthotics and Prosthetics User's Survey (OPUS) at 4 months post-intervention. | 2 weeks pre-intervention; baseline; 1 month post-intervention; 4 months post-intervention
  The CSD contains 9 items rated on a 5-point Likert scale ranging from 0 ('strongly disagree') to 4 ('strongly agree), with a total score ranging from 0-36. Since the CSD is not yet available in Dutch, the investigators will translate it into the Dutch language and assess its content validity, structural validity, and reliability in Dutch orthotic users.
Change from baseline in satisfaction assessed with the Dutch version of the Quebec User Evaluation of Satisfaction with Assistive Technology (D-QUEST) at 4 months post-intervention | Baseline; 1 month post-intervention; 4 months post-intervention
  The D-QUEST assesses satisfaction with aspects related to the device and provided services. For this study, only the device-part of the D-QUEST will be used, which comprises 8 questions about certain characteristics of the orthotic device, all scored on a 5-point scale (from 'not satisfied at all' to 'very satisfied'), with a total score ranging from 8-40 (with 40 being the best possible satisfaction score).
Change in quality of life on the 5-dimension 5-level EuroQol (EQ-5D-5L) at 4 months post-intervention. | Baseline; 1 month post-intervention, 4 months post-intervention
  The EQ-5D-5L contains five questions about mobility, self-care, usual activities, pain/discomfort, and anxiety and depression scored on a 5-point scale indicating the degree of problems with each dimension and one question about experienced health scored on a 0-100 visual analogue scale.
Production time of the orthosis (in minutes). | From start of the intervention up to delivery of the orthosis
  For each step in manufacturing the orthosis until final delivery, time will be recorded (with a stopwatch).
Production costs of the orthosis (in euro). | From start of the intervention up to delivery of the orthosis
  Costs of the conventional orthoses will be retrospectively inventoried from the administration records of OIM. Costs related to the manufacturing of the 3D-printed orthoses will be prospectively assessed.
Change from baseline in personal goals at 4 month post-intervention. | Baseline; 1 month post-intervention, 4 months post-intervention
  An in-house usability questionnaire will be used to inventory information on personal goals of the orthosis, and whether this goal has been achieved (scored on a 10-point-scale, ranging from 1: not achieved at all to 10: very well achieved).
Change from baseline in orthosis use at 4 month post-intervention. | Baseline; 1 month post-intervention, 4 months post-intervention
  An in-house usability questionnaire will be used to inventory how often the orthosis is used, classified in 5 categories; ranging from never until 6-7 days a week.
Patient and therapist experiences with the 3D orthosis | 1 month post-treatment
  Experiences of patients and health care providers with respect to the time window of the 3D intervention and satisfaction with the treatment process will be assessed with an in-house questionnaire, with items scored on a 5-point Likert scale.
Number of visits for fabrication of the 3D orthosis | From start of the intervention up to delivery of the orthosis
  The total number of visits for fabricating the 3D orthosis will be obtained from the administration records of OIM

OTHER OUTCOMES:
Adverse events | up to 4 months post intervention
  The following adverse events reported by the participant or observed by the investigator or orthotist will be recorded; pressure sores, abrasions, pain due to the orthosis, and material damage of the orthosis.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. Frans Nollet, MD PhD, Study Director — Amsterdam UMC, location AMC
Locations (1):
- Department of rehabilitation medicine Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) and meta data will be made available to third parties via Figshare. Other anonymized IPD and documents will be made available on request including data analysis codes such as SPSS syntaxes or R scripts.

REFERENCES:
- [Background] Oud TAM, Lazzari E, Gijsbers HJH, Gobbo M, Nollet F, Brehm MA. Effectiveness of 3D-printed orthoses for traumatic and chronic hand conditions: A scoping review. PLoS One. 2021 Nov 18;16(11):e0260271. doi: 10.1371/journal.pone.0260271. eCollection 2021. PMID 34793566
- [Background] Oud T, Kerkum Y, de Groot P, Gijsbers H, Nollet F, Brehm MA. Production Time and User Satisfaction of 3-Dimensional Printed Orthoses For Chronic Hand Conditions Compared With Conventional Orthoses: A Prospective Case Series. J Rehabil Med Clin Commun. 2021 Feb 12;4:1000048. doi: 10.2340/20030711-1000048. eCollection 2021. PMID 33884150
- [Derived] Oud T, Tuijtelaars J, Schenk J, Nollet F, Brehm MA. Validity and reliability of the Dutch translation of the OPUS' client satisfaction with device module in chronic users of hand orthoses. Health Qual Life Outcomes. 2023 Aug 21;21(1):93. doi: 10.1186/s12955-023-02181-3. PMID 37605151
- [Derived] Oud T, Tuijtelaars J, Bogaards H, Nollet F, Brehm MA. Preliminary effectiveness of 3D-printed orthoses in chronic hand conditions: study protocol for a non-randomised interventional feasibility study. BMJ Open. 2023 Apr 6;13(4):e069424. doi: 10.1136/bmjopen-2022-069424. PMID 37024252